CLINICAL TRIAL: NCT03900949
Title: A Phase I Study to Evaluate the Safety and Tolerability of Gemtuzumab Ozogamicin and Midostaurin When Used in Combination With Standard Cytarabine and Daunorubicin Induction for Newly Diagnosed FLT3-mutated Acute Myeloid Leukemia
Brief Title: Gentuzumab Ozogamicin and Midostaurin Combination With Standard Cytarabine and Danunorubi Midostaurin as a Novel Approach to Treating Patients With Newly Diagnosed FLT-3 Mutated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uma Borate (Other)
Responsible Party: Sponsor-Investigator, Uma Borate, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21190; NCI-2019-01726 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: FLT; FLT-3; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Stem Cell Transplantation; Cytarabine; Daunorubicin; Gemtuzumab; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (gemtuzumab ozogamicin, cytarabine, daunorubicin) (Experimental): INDUCTION THERAPY: Cytarabine intravenously (IV) on days 1-7, daunorubicin IV on days 1-3 and midostaurin 50 mg orally (PO) twice daily (BID) on days 8-21. Gemtuzumab ozogamicin IV may be given either on days 1, or days 1 and 4 or days 1, 4 and 7. RE-INDUCTION THERAPY: Between days 14 and 21 of Induction Therapy, patients may receive a single 28-day cycle of cytarabine and daunorubicin with or without midostaurin per the treating physician. Patients may also undergo allogeneic stem cell transplantation (SCT) or receive consolidation therapy. CONSOLIDATION THERAPY: PATIENTS < 60 YEARS: high dose cytarabine (HiDAC) IV on days 1, 3, and 5 and gemtuzumab ozogamicin IV on day 1 of cycle 1 and midostaurin 50 mg PO BID on days 8-21. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. PATIENTS >= 60 YEARS: Same as above except cytarabine (MiDAC) IV on days 1, 3, and 5.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Gemtuzumab Ozogamicin; Drug: Midostaurin

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic SCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Drug: Midostaurin — Given PO
  Other Names: CGP 41251; CGP41251; N-Benzoyl-Staurosporine; N-Benzoylstaurosporine; PKC-412; PKC412; Rydapt

SUMMARY:
This phase I study hopes to explore how safe and tolerable is the combination of gemtuzumab ozogamicin (GO) and midostaurin, with the standard induction therapy (cytarabine and daunorubicin) in patients with newly diagnosed FLT-3 mutated Acute Myeloid Leukemia (AML). GO is FDA approved for the treatment of adults with newly diagnosed CD33 positive AML and used in combination with chemotherapy, cytarabine and daunorubicin. Midostaurin is FDA approved for use with cytarabine and daunorubicin in patients with FLT3-mutated AML. By combining standard induction therapy with GO and midostaurin, our aim is to investigate a novel approach to treating patients with newly diagnosed FLT3-mutated AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the maximum tolerated dose (MTD) of combining gemtuzumab ozogamicin (GO) to the induction regimen of cytarabine and daunorubicin (DA) and midostaurin.

SECONDARY OBJECTIVES:

I. To assess the frequency of early death associated with study treatment. II. To evaluate the preliminary efficacy of the study treatment. III. To assess the safety profile of the study treatment.

EXPLORATORY OBJECTIVES:

I. Quantify CD33 expression on acute myeloid leukemia (AML) blasts. II. Determine the CD33 single-nucleotide polymorphism (SNP) status previously reported to correlate with response and correlate clinical outcomes of patients with the CD33 genotype.

OUTLINE: This is a dose finding study to identify the maximum tolerated dose (MTD) schedule of GO, and its safety and tolerability in combination with midostaurin in FLT3-mutated newly diagnosed AML patients.

INDUCTION THERAPY: Patients receive cytarabine intravenously (IV) on days 1-7, daunorubicin IV on days 1-3 and midostaurin 50mg orally (PO) twice daily (BID) on days 8-21. Patients also receive gemtuzumab ozogamicin IV either on day or days 1 and 4 or days 1, 4 and 7 depending on dose level in the absence of disease progression or unacceptable toxicity.

RE-INDUCTION THERAPY: Between days 14 and 21 of Induction Therapy, patients who achieve at least 5% bone marrow blasts after an optional bone marrow biopsy may receive a single 28-day cycle of cytarabine and daunorubicin with or without midostaurin per the treating physician. Patients who achieve a complete remission (CR) or complete remission with incomplete blood count recovery (CRi) may undergo allogeneic stem cell transplantation (SCT) or receive consolidation therapy.

CONSOLIDATION THERAPY:

PATIENTS < 60 YEARS: Patients receive high dose cytarabine (HiDAC) IV on days 1, 3, and 5 and gemtuzumab ozogamicin IV on day 1 of cycle 1 and midostaurin 50mg PO BID on days 8-21. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

PATIENTS >= 60 YEARS: Patients receive cytarabine (MiDAC) IV on days 1, 3, and 5 and gemtuzumab ozogamicin IV on day 1 of cycle 1 and midostaurin 50mg PO BID on days 8-21. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Newly diagnosed AML as confirmed by bone marrow and/or peripheral blood examination as indicated, with:

  * Confirmed CD33 positivity, per institutional standards
  * Presence of FLT3 internal tandem duplication (ITD) or tyrosine kinase domain (TKD) mutation as confirmed by next-generation sequencing (NGS) or other molecular method
* Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN; local laboratory)
* Alanine aminotransferase (ALT) < 2.5 x ULN
* Total bilirubin < 2 x ULN (except for patients with known Gilbert's syndrome)
* Calculated creatinine clearance (according to the Cockcroft-Gault equation) > 40 mL/min OR serum creatinine < 1.5 x the ULN
* Female patients of childbearing potential must agree to use adequate contraception (2 forms of contraception or abstinence) from the screening visit until 6 months following the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Male patients of childbearing potential having intercourse with females of childbearing potential must agree to abstain from heterosexual intercourse or have their partner use 2 forms of contraception from the screening visit until 4 months following the last dose of study treatment. They must also refrain from sperm donation from the screening visit until 4 months following the last dose of study treatment

Exclusion Criteria:

* Isolated myeloid sarcoma (meaning, patients must have blood or marrow involvement to enter study)
* Acute promyelocytic leukemia (per World Health Organization classification)
* Active central nervous system (CNS) involvement by AML, as assessed at discretion of principal investigator (PI) or treating physician and confirmed by lumbar puncture
* Except for hydroxyurea, no other prior systemic anti-AML therapies may have been received prior to starting study therapy
* Known history of veno-occlusive disease
* Known active human immunodeficiency virus (HIV), active hepatitis B or active hepatitis C infection
* Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III or IV heart failure, severe uncontrolled ventricular arrhythmias
* Patients with uncontrolled infection will not be enrolled until infection is treated
* Any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol
* Inability to take oral medication
* Hypersensitivity to any study agent, or its excipients, when administered alone
* Pregnancy or breastfeeding at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of combining gemtuzumab ozogamicin with cytarabine, daunorubicin, and midostaurin | 42 days after start of last induction (i.e. induction or re-induction)
  The MTD will be estimated using isotonic regression. An incidence of dose limiting toxicity at each dose level will be summarized.

SECONDARY OUTCOMES:
Incidence of 30-day treatment-related mortality | Up to 30 days after receiving initial induction therapy
  Will be estimated with exact confidence intervals.
Rate of complete composite remission (CCR) | At end of consolidation treatment (up to 120 days)
  Complete composite remission is defined as meeting criteria for complete remission (CR), complete remission with incomplete blood count recovery (CRi), or complete remission with incomplete platelet recovery (CRp). Will be measured and reported with 95% exact confidence intervals.
Objective response rate (ORR) | At end of consolidation treatment (up to 120 days)
  ORR is defined as the sum of CR, CRi, Morphologic leukemia-free state (MLFS), and Partial remission (PR). Will be measured and reported with 95% exact confidence intervals.
Event free survival | From date of primary refractory disease, or relapse from complete response (CR) or complete remission with incomplete blood count recovery (CRi) , or death from any cause, assessed up to 24 months
  EFS will be measured from start of on-study therapy (i.e., Day 1) to the date of primary refractory disease, relapse from CR or CRi, or death from any cause. Participants not known to have failed induction therapy, relapsed, or died at time of last follow-up will be censored on the date they were last examined (i.e., 2 years following completion of on-study therapy). The Kaplan-Meier method will be used. Mean and/or median survival and 95% confidence intervals will be reported, if available.
Duration of response | From date of first documented response (CR, CRi) to date of documented relapse, assessed up to 24 months
  For only participants that achieve CR or CRi, the DoR is measured from the date of first documented response (CR, CRi) until the date of relapse. Participants not known to have relapsed at time of last follow-up will be censored on the date they were last examined (i.e., 2 years following completion of on-study therapy). The Kaplan-Meier method will be used. Mean and/or median survival and 95% confidence intervals will be reported, if available.
Relapse-free survival | From date of first documented response (CR, CRi) to date of relapse or death from any cause, assessed up to 24 months
  For only participants that achieve CR or CRi, RFS will be measured from the date of first documented response (CR, CRi) to the date of relapse or death from any cause. Participants not known to have relapsed or died at time of last follow-up will be censored on the date they were last examined (i.e., 2 years following completion of on-study therapy). The Kaplan-Meier method will be used. Mean and/or median survival and 95% confidence intervals will be reported, if available.
Overall survival | From start of treatment until death, assessed up to 24 months
  The Kaplan-Meier method will be used. Mean and/or median survival and 95% confidence intervals will be reported, if available.
Incidence of adverse events and serious adverse events | Up to 90 days after last dose of treatment
  Will be tabulated and summarized by severity and major organ site according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
CD33 expression | Up to 24 months
  Will be summarized descriptively. CD33 expression will be correlated with CCR and ORR using Fisher's exact test and with time-to-event endpoints using a log-rank test.
CD33 single nucleotide polymorphism (SNP) | Up to 24 months
  Will be summarized descriptively. The presence/absence of CD33 SNPs will be correlated with CCR and ORR using Fisher's exact test and with time-to-event endpoints using a log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Uma Borate, M.D., Principal Investigator — The Ohio State Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University Knight Cancer Institute - Northwest Portland, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jain J, Pugh K, Handa S, Dvorak-Kornaus KM, Zhao Q, Walter RB, Cook R, Saultz J, Swords R, Li J, Laszlo GS, Grieselhuber NR, Mims AS, Larkin KTM, Sahasrabudhe K, Blachly JS, Behbehani GK, Eisfeld AK, Long M, Srisuwananukorn A, Koenig KL, Borate U. Safety of gemtuzumab ozogamicin with cytarabine, daunorubicin, and midostaurin induction in FLT3-mutated AML. Blood Neoplasia. 2025 Oct 9;3(1):100171. doi: 10.1016/j.bneo.2025.100171. eCollection 2026 Feb. PMID 41488889
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2024-07-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT03900949/ICF_000.pdf